CLINICAL TRIAL: NCT02854618
Title: Study of the Immune Response T Anti-tumoral Cluster of Differentiation 4 (CD4) for Patients Treated for a Metastatic Breast Cancer by Everolimus Within the Framework of Its Marketing Authorization
Brief Title: Immune Response for Patients With Metastatic Breast Cancer Treated by Everolimus
Acronym: EVERIMMUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P/2012/159
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus treatment (Experimental)
  Interventions: Other: additional blood sample

INTERVENTIONS:
Other: additional blood sample

SUMMARY:
This study evaluates the immune response for patients affected by metastatic breast cancer treated by everolimus

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for a treatment by everolimus in association with the exemestane
* Performance status of 0,1 or 2 according to the WHO
* Patients affected of a breast cancer advanced and\or metastatic HER2 negative expressing the hormonal receptor RH +
* menopausal Patients

Exclusion Criteria:

* Psychiatric disease compromising the understanding of the information or the realization of the study
* Vulnerable people according to the law (minors, adults under protection, private persons of freedom)
* Histories of cancer in 5 years preceding the diagnosis (except breast cancer, squamous-cell)
* Not menopausal women
* Unaffiliated people to the Social Security
* People being for the period of exclusion from another study
* Hypersensitivity in the active substance, in the other by-products of the rapamycin or in one of the excipients.
* Symptomatic visceral achievement
* Legal incapacity or limited legal capacity

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-11-26 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
level of the spontaneous anti-telomerase response | 12 months
  evaluation by Enzyme-Linked Immunospot (ELIspot) and by Enzyme-Linked Immunosorbent Assay (ELISA test)

SECONDARY OUTCOMES:
T lymphocytes level | 12 months
everolimus level in serum patients | 12 months
angiopoietin 2 level | 12 months
CD138 level | 12 months
ps6K expression | 12 months
Merlin expression | 12 months
neuropilin 2 expression | 12 months
quality of life | 12 months
  EUROQOL EQ-5D, EORTC QLQ-C30 and BR 23

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No